CLINICAL TRIAL: NCT01052519
Title: Intraoperative Goal-directed Fluid Management in Non-Obese and Obese Patients Undergoing Laparoscopic Surgery
Brief Title: Obesity and Goal-directed Intraoperative Fluid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Kabon, PD. MD., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 708/2009, local IRB
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: Obesity; Esophageal Doppler monitoring; tissue oxygen tension
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- obese control (No Intervention)
- obese goal-directed (Active Comparator)
  Interventions: Other: Goal directed fluid therapy
- non-obese goal directed (Active Comparator)
  Interventions: Other: Goal directed fluid therapy

INTERVENTIONS:
Other: Goal directed fluid therapy — Fluid will be administered to reach maximal stroke volume during the intraoperative period.
  Arms: non-obese goal directed; obese goal-directed

SUMMARY:
The purpose of the study is to compare non-obese patients (BMI≤ 30 kg/m2)versus obese patients (BMI> 30 kg/m2) in regard of their respective needs for intraoperative fluid therapy during laparoscopic surgery.

Specifically the investigators will test the hypothesis that subcutaneous tissue oxygenation (PsqO2)is increased in obese patients when fluid management is optimized by means of esophageal Doppler monitoring compared to obese patients undergoing standard fluid management.

Furthermore the investigators will test the hypothesis that PsqO2 is decreased in obese patients undergoing conventional fluid therapy compared to non-obese patients when fluid management is optimized. Thus the investigators assume that PsqO2 is similar in obese and non-obese patients when fluid management is optimized in both groups.

DETAILED DESCRIPTION:
Hemodynamic stability and normovolemia are critical determinants of tissue perfusion and oxygenation. Adequate tissue oxygenation is essential to maintain normal physiologic functions and to reduce complications, such as wound infections.

Fat tissue is relatively hypoperfused and, therefore, poorly oxygenated. Subcutaneous tissue oxygenation in the obese is thus critically low and even supplemental oxygen only slightly increases subcutaneous oxygenation.It is likely that poor subcutaneous oxygenation in the obese surgical patients results in part from inadequate intraoperative fluid replacement.

It remains unknown how to hydrate obese surgical patients best. The most physiologic approach for perioperative fluid replacement is now thought to be goal-directed management, using stroke volume as the treatment parameter.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (BMI≤ 30kg/m2) and obese patients (BMI > 30 kg/m2)
* undergoing laparoscopic elective fundoplication or elective bariatric surgery

Exclusion Criteria:

* decompensate heart failure
* documented coronary artery disease
* renal insufficiency
* severe chronic obstructive pulmonary disease
* symptoms of infection or sepsis
* esophageal disease (excepting gastro-esophageal reflux without any other esophageal alteration).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Subcutaneous tissue oxygenation | intraoperative and 2 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kabon, MD, Principal Investigator — MUW
Locations (1):
- Department of Anesthesiology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Kabon B, Nagele A, Reddy D, Eagon C, Fleshman JW, Sessler DI, Kurz A. Obesity decreases perioperative tissue oxygenation. Anesthesiology. 2004 Feb;100(2):274-80. doi: 10.1097/00000542-200402000-00015. PMID 14739800
- [Background] Fleischmann E, Kurz A, Niedermayr M, Schebesta K, Kimberger O, Sessler DI, Kabon B, Prager G. Tissue oxygenation in obese and non-obese patients during laparoscopy. Obes Surg. 2005 Jun-Jul;15(6):813-9. doi: 10.1381/0960892054222867. PMID 15978153
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Derived] Muhlbacher J, Luf F, Zotti O, Herkner H, Fleischmann E, Kabon B. Effect of Intraoperative Goal-Directed Fluid Management on Tissue Oxygen Tension in Obese Patients: a Randomized Controlled Trial. Obes Surg. 2021 Mar;31(3):1129-1138. doi: 10.1007/s11695-020-05106-x. Epub 2020 Nov 27. PMID 33244655